CLINICAL TRIAL: NCT01853124
Title: Impact of Emergency Department Probiotic Treatment of Pediatric Gastroenteritis: Randomized Controlled Trial
Brief Title: Emergency Department Probiotic Treatment of Pediatric Gastroenteritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dr. Stephen Freedman (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Alberta Children's Hospital (Other); The Hospital for Sick Children (Other); Children's Hospital of Eastern Ontario (Other); St. Justine's Hospital (Other); IWK Health Centre (Other); Institut Rosell Lallemand (Industry); London Health Sciences Center, Children's Hospital (Unknown)
Responsible Party: Sponsor-Investigator, Dr. Stephen Freedman, Associate Professor of Pediatrics; Alberta Children's Hospital Foundation Professor in Child Health and Wellness Alberta Children's Hospital Theme Lead, University of Calgary
Organization: University of Calgary (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: REB13-0045
Record Dates: First submitted 2013-05-09; First posted 2013-05-14 (Estimated); Last update posted 2018-03-02 (Actual); Status verified 2018-02

CONDITIONS: Gastroenteritis
Keywords: Diarrhea
MeSH Terms: conditions — Gastroenteritis; Diarrhea

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lacidofil (Experimental): Lacidofil sachet containing active ingredients
  Interventions: Drug: Lacidofil
- Placebo (Placebo Comparator): Placebo sachet containing inactive ingredients
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — All patients in this arm of the study will take 1 sachet containing inactive ingredients (maltodextrin, magnesium stearate, and ascorbic acid) twice daily for 5 days. Doses should be ideally separated by 12 hours (minimum of 8 hours) and taken within 30 minutes of food/drink. If the child vomits within 15 minutes of medication administration (initial or subsequent dose), the dose will be repeated. Total of 2 sachets per day for 5 days.
  Arms: Placebo
Drug: Lacidofil — All patients in this arm of the study will take 1 sachet twice daily for 5 days. Each sachet will contain a minimum of 4 billion colony-forming units (CFU) of Lactobacillus rhamnosus Rosell-11 (95%) and L. helveticus Rosell-52 (5%). The total weight of all ingredients is 1 gm. Doses should be ideally separated by 12 hours (minimum of 8 hours) and taken within 30 minutes of food/drink. If the child vomits within 15 minutes of medication administration (initial or subsequent dose), the dose will be repeated. Total daily dose = 8 billion CFU x 5 days.
  Arms: Lacidofil

SUMMARY:
The objective of this study is to determine for previously healthy children who present to a Canadian Emergency Department (ED) with acute gastroenteritis (infection or irritation of the digestive tract); if compared with placebo, the administration of a probiotic agent (Lacidofil) will result in a significantly lower proportion of children developing moderate to severe disease over the subsequent 2 weeks and will not be associated with a significantly greater occurrence of side effects.

DETAILED DESCRIPTION:
The burden of acute gastroenteritis (AGE) on children and their families continues to be enormous. It accounts for 1.7 million pediatric emergency department (ED) visits annually in the United States and nearly 240,000 in Canada. Children often suffer from prolonged and severe illness; amongst hospitalized Canadian children, 19% have clinical sepsis, 7% seizures and 4% require intensive care unit admission.3 In a study that we conducted at 11 Canadian EDs, 51% of children experienced moderate to severe disease. Parents rate such episodes as being equivalent to a 10 day admission (moderate) and persistent moderate hearing loss (severe). The burden is augmented by the 50% household transmission rate2, 6 and 42% prolonged work absenteeism rate. Apart from supportive care, health-care providers have little to offer to relieve suffering.

Probiotics, which are defined as viable microbial preparations that have a beneficial effect on the health of the host, represent a rapidly expanding field. While they are available as over-the-counter products, according to the National Institutes of Health, the Food and Drug Administration has not yet approved a single agent for any health claims. Further, a 2012 meta-analysis concluded that there is limited data to support their indications and no published pediatric gastroenteritis trials reported on side effects. Thus, understanding the benefits and side effects of probiotics is crucial before widespread use can be endorsed. Although probiotic clinical trials have been performed, only one (still unpublished) has been ED based. Most studies to date have been significantly flawed and guidelines do NOT endorse their use stating that well-controlled human trials are needed. Consequently, we and others have found that they are rarely used in clinical practice. Reasons cited include (1) questionable clinical meaning to the outcomes evaluated thus far; (2) absence of studies in the appropriate patient population, and (3) a lack of confidence in the quality of probiotic agents studied.

This study will address (1) the needs of the medical community, which is aware of the widening gap between the number of important pediatric and adult trials and (2) the interest of caregivers in "probiotics" - 71% are aware of the term; 31% believe they may be beneficial in children with diarrhea, and > 90% would administer a probiotic if it could make their child better. Furthermore, our pilot study has provided promising preliminary data and has proven the feasibility of our methods. Thus we are poised to conduct a randomized controlled trial (RCT)that will definitively determine if meaningful benefits are derived from probiotic use and will provide critical information regarding their mechanism of action. This information will impact on practice, the burden of disease, and ensure that children receive the best care possible. The results of our proposed RCT will enable guidelines to either clearly endorse or recommend against the routine use of a probiotic agent in children with Acute Gastroenteritis.

We also hypothesize that the therapeutic benefits of probiotics in children with AGE vary by infecting pathogen. We have assembled a team to bridge the gap between the clinical RCT team, molecular diagnostics, and immunologic to quantify the pathogen-specific effects of probiotics. The latter is likely because there are distinct mechanisms (e.g. invasive, inflammatory, non-inflammatory) by which pathogens cause clinical symptoms. Similarly, probiotic effects are exerted through multiple modes-of-action (e.g. direct antimicrobial activity, competitive exclusion, immune response stimulation, inhibition of virulence gene or protein expression). The simultaneous evaluation of pathogen-specific effects on clinical, microbiological and immunological levels has not previously been performed.

The knowledge gained through this multi-faceted approach will inform understanding of the probiotic-host-pathogen interactions that are responsible for improved clinical outcomes in children with AGE. Our study population, outpatient children, is both the main group of patients who suffer from AGE as well as the main consumer of probiotics. Thus, our findings will be relevant and ready for translation into clinical care while simultaneously opening up avenues for future research.

The principal questions to be addressed are as follows:

Hypotheses: In children aged 3-48 months presenting to an ED with less than 72 hours of AGE like symptoms, compared with placebo, the administration of a probiotic agent:

1. Will result in a significantly lower proportion of children developing moderate to severe disease over the subsequent 2 weeks.
2. Will not be associated with a significantly greater occurrence of minor side effects.
3. Will be associated with a greater increase in secretory IgA (sIgA).
4. Will have varying effects based on the etiologic pathogen, given the diverse underlying pathophysiologic processes induced by the causative agents and the multiple mechanisms of action of probiotics.

Clinical Efficacy:

Primary Question: For previously healthy children, ages 3-48 months, who present to an ED with less than 72 hours of AGE like symptoms, is the proportion who develop moderate to severe disease [Modified Vesikari Score (MVS) ≥ 9] following ED evaluation, significantly different in those who receive a probiotic agent (Lacidofil) compared to those who receive placebo?

Secondary Questions: In this group of patients, amongst those receiving active treatment versus placebo:

1. Is there a difference in the (a) duration of diarrhea or (b) duration of vomiting?
2. Is there a difference in the proportion who require an unscheduled health care provider visit?
3. Is there a difference in the effectiveness of treatment based on the infecting pathogen?

Side Effect Profile:

Question: In this group of patients, is the proportion that experiences a side effect (e.g. bloating, fever, abdominal distention, rash) significantly different in those who receive Lacidofil compared to placebo?

Mechanism of Action:

Question: In this group of patients, are fecal sIgA levels 5 days and 4 weeks after the initiation of treatment higher in those who receive Lacidofil compared to those who receive placebo?

Microbiologic - Stool Pathogen-Specific Load:

Question: In this group of patients, is there a difference in the pathogen specific reduction in stool pathogen load in those who receive Lacidofil compared to those who receive placebo?

ELIGIBILITY:
Inclusion Criteria:

* Presence of diarrhea: defined as ≥ 3 watery stools in a 24-hour period
* Duration of vomiting and/or diarrhea < 72 hours
* Age 3 to < 48 months

Exclusion Criteria:

* Presence of an indwelling vascular access line or structural heart disease
* Taking immunosuppressive therapy, or known history of immunodeficiency
* Hematochezia in the preceding 72 hours, underlying significant chronic gastrointestinal problem or inflammatory bowel disease
* Family member with an indwelling vascular access line, on immunosuppressive therapy, or with a known immunodeficiency
* Bilious vomiting
* Probiotic use (supplement) in the preceding 2 weeks
* Previously enrolled in this trial
* Daily follow-up not possible
* Allergy to Soy
* Pre-existing (known) pancreatic dysfunction or insufficiency
* Oral or Gastrointestinal surgery within preceding 7 days

Ages: 3 Months to 48 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 886 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Development of moderate to severe disease in the 2 weeks after the index visit | Measured daily for 14 days

SECONDARY OUTCOMES:
Duration of Diarrhea | Daily for 14 days
Duration of Vomiting | Daily for 14 days
Return visits for unscheduled care to a health care provider related to vomiting, diarrhea, dehydration, fever, or fluid refusal, within two weeks | Daily for 14 days
Work and Daycare Absenteeism | Daily for 14 days

OTHER OUTCOMES:
Side Effect Profile | Daily for 14 days
  Determine if short course probiotic administration to young children with acute gastroenteritis is associated with an increase in minor side effects
Mechanism of Action | 28 Days
  Determine if probiotic administration increases fecal secretory IgA levels in children with acute gastroenteritis
Pathogen Load Quantification | Determine if a 5-day probiotic treatment course administered to children with acute gastroenteritis results in pathogen-specific reductions in stool pathogen load
  5 Days

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Freedman, MD, Principal Investigator — University of Calgary
Locations (6):
- Canada (6):
  - Alberta Children's Hospital, Calgary, Alberta
  - IWK Health Centre, Halifax, Nova Scotia
  - Children's Hospital, London Health Sciences Center, London, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - The Hospital for Sick Children, Toronto, Ontario
  - Centre Hospitalier Universitaire Sainte Justine, Montreal, Quebec

REFERENCES:
- [Derived] Horne RG, Freedman SB, Johnson-Henry KC, Pang XL, Lee BE, Farion KJ, Gouin S, Schuh S, Poonai N, Hurley KF, Finkelstein Y, Xie J, Williamson-Urquhart S, Chui L, Rossi L, Surette MG, Sherman PM. Intestinal Microbial Composition of Children in a Randomized Controlled Trial of Probiotics to Treat Acute Gastroenteritis. Front Cell Infect Microbiol. 2022 Jun 14;12:883163. doi: 10.3389/fcimb.2022.883163. eCollection 2022. PMID 35774405
- [Derived] Freedman SB, Finkelstein Y, Pang XL, Chui L, Tarr PI, VanBuren JM, Olsen C, Lee BE, Hall-Moore CA, Sapien R, O'Connell K, Levine AC, Poonai N, Roskind C, Schuh S, Rogers A, Bhatt S, Gouin S, Mahajan P, Vance C, Hurley K, Powell EC, Farion KJ, Schnadower D. Pathogen-Specific Effects of Probiotics in Children With Acute Gastroenteritis Seeking Emergency Care: A Randomized Trial. Clin Infect Dis. 2022 Aug 24;75(1):55-64. doi: 10.1093/cid/ciab876. PMID 34596225
- [Derived] Freedman SB, Horne R, Johnson-Henry K, Xie J, Williamson-Urquhart S, Chui L, Pang XL, Lee B, Schuh S, Finkelstein Y, Gouin S, Farion KJ, Poonai N, Hurley K, Schnadower D, Sherman PM; Pediatric Emergency Research Canada Probiotic Regimen for Outpatient Gastroenteritis Utility of Treatment (PROGUT) Trial Group. Probiotic stool secretory immunoglobulin A modulation in children with gastroenteritis: a randomized clinical trial. Am J Clin Nutr. 2021 Apr 6;113(4):905-914. doi: 10.1093/ajcn/nqaa369. PMID 34269370
- [Derived] Freedman SB, Roskind CG, Schuh S, VanBuren JM, Norris JG, Tarr PI, Hurley K, Levine AC, Rogers A, Bhatt S, Gouin S, Mahajan P, Vance C, Powell EC, Farion KJ, Sapien R, O'Connell K, Poonai N, Schnadower D; Pediatric Emergency Research Canada and Pediatric Emergency Care Applied Research Networks. Comparing Pediatric Gastroenteritis Emergency Department Care in Canada and the United States. Pediatrics. 2021 Jun;147(6):e2020030890. doi: 10.1542/peds.2020-030890. Epub 2021 May 20. PMID 34016656
- [Derived] Poonai N, Powell EC, Schnadower D, Casper TC, Roskind CG, Olsen CS, Tarr PI, Mahajan P, Rogers AJ, Schuh S, Hurley KF, Gouin S, Vance C, Farion KJ, Sapien RE, O'Connell KJ, Levine AC, Bhatt S, Freedman SB; Pediatric Emergency Care Applied Research Network (PECARN) and Pediatric Emergency Research Canada (PERC). Variables Associated With Intravenous Rehydration and Hospitalization in Children With Acute Gastroenteritis: A Secondary Analysis of 2 Randomized Clinical Trials. JAMA Netw Open. 2021 Apr 1;4(4):e216433. doi: 10.1001/jamanetworkopen.2021.6433. PMID 33871616
- [Derived] Freedman SB, Williamson-Urquhart S, Farion KJ, Gouin S, Willan AR, Poonai N, Hurley K, Sherman PM, Finkelstein Y, Lee BE, Pang XL, Chui L, Schnadower D, Xie J, Gorelick M, Schuh S; PERC PROGUT Trial Group. Multicenter Trial of a Combination Probiotic for Children with Gastroenteritis. N Engl J Med. 2018 Nov 22;379(21):2015-2026. doi: 10.1056/NEJMoa1802597. PMID 30462939
- [Derived] Freedman SB, Williamson-Urquhart S, Schuh S, Sherman PM, Farion KJ, Gouin S, Willan AR, Goeree R, Johnson DW, Black K, Schnadower D, Gorelick MH; Pediatric Emergency Research Canada (PERC) Gastroenteritis Study Group. Impact of emergency department probiotic treatment of pediatric gastroenteritis: study protocol for the PROGUT (Probiotic Regimen for Outpatient Gastroenteritis Utility of Treatment) randomized controlled trial. Trials. 2014 May 14;15:170. doi: 10.1186/1745-6215-15-170. PMID 24885220